CLINICAL TRIAL: NCT03258528
Title: Effect of Right Lateral Position With Head Elevation on Tracheal Aspirate Pepsin in Ventilated Preterm Neonates: Randomized Controlled Trial
Brief Title: Effect of Right Lateral Position on Ventilated Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Mohamed Shinkar, Prinicpal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Neonatal Reflux
Record Dates: First submitted 2017-08-18; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- right lateral position group (Active Comparator): Neonates kept in the right lateral position for 6 hours with head tilted 30 degree upward with rolled towel supports the infant back at 90 degree angle on the bed.
  Interventions: Behavioral: positioning
- supine position group (Active Comparator): Neonates kept in supine position for 6 hours with head tilted 30 degrees upward.
  Infants were fed while in their positions via feeding tube.
  Interventions: Behavioral: positioning

INTERVENTIONS:
Behavioral: positioning — Positioning neonates for 6 hours either in right lateral position or supine position

SUMMARY:
Objective: to evaluate the effect of right lateral positioning in comparison with supine positioning on tracheal aspirate pepsin levels as a marker of aspiration of gastric contents in ventilated preterm neonates. Study design: This randomized controlled trial was conducted on 60 ventilated preterm neonates < 35 weeks. They were randomized into 2 groups; one group composed of 30 neonates that were nursed in right lateral position for 6 hours while the other group composed of 30 neonates that were nursed in supine position for 6 hours. Tracheal aspirate sample was obtained from each neonate in both groups just after the end of 6 hours and pepsin level was measured.

DETAILED DESCRIPTION:
Objective: to evaluate the effect of right lateral positioning in comparison with supine positioning on tracheal aspirate pepsin levels as a marker of aspiration of gastric contents in ventilated preterm neonates. Study design: This randomized controlled trial was conducted on 60 ventilated preterm neonates < 35 weeks. They were randomized into 2 groups; one group composed of 30 neonates that were nursed in right lateral position for 6 hours while the other group composed of 30 neonates that were nursed in supine position for 6 hours. Tracheal aspirate sample was obtained from each neonate in both groups just after the end of 6 hours and pepsin level was measured. Ventilatory settings were observed before and during the intervention and neonates were followed up for development of bronchopulmpnary dysplasia (BPD).

ELIGIBILITY:
Inclusion Criteria:

* A total of 60 preterm neonates < 35 weeks gestational age were enrolled in the study, Inclusion criteria were tracheal intubated mechanically ventilated neonates for more than 72 hours, feeding >30ml/kg/day via nasogastric tube.

Exclusion Criteria:

* Neonates with perinatal asphyxia, intracranial hemorrhage grade 3 or 4, periventricular leukomalacia, major congenital anomalies, gastrointestinal anomalies such as tracheoesophageal fistula, or necrotizing enterocolitis , receiving xanthine derivatives, H2 blockers, prokinetics, proton pump inhibitors or sedatives were excluded.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
tracheal aspirate pepsin | 6 hours
  Tracheal aspirate sample was obtained from each neonate in both groups just after the end of 6 hours and pepsin level was measured

IPD SHARING:
Plan to Share IPD: Undecided